CLINICAL TRIAL: NCT00831532
Title: A Phase 1, Non-Randomized, Open-Label, Single-Dose Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Dimebon [Pf-01913539] In Subjects With Hepatic Impairment And Normal Hepatic Function
Brief Title: Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Dimebon [Pf-01913539] In Subjects With Hepatic Impairment And Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1451018
Record Dates: First submitted 2009-01-20; First posted 2009-01-29 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Hepatic Failure
Keywords: Dimebon Hepatic Impairment
MeSH Terms: conditions — Liver Failure | interventions — latrepirdine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal (Experimental): Healthy Volunteers
  Interventions: Drug: Dimebon
- Mild Hepatic Impairment (Experimental): Mild hepatic impairment patients
  Interventions: Drug: Dimebon
- Moderate hepatic Impairment (Experimental): Moderate Hepatic Impairment Patients
  Interventions: Drug: Dimebon
- Severe Hepatic Impairment (Experimental): Severe Hepatic Impairment Patients
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — Dimebon 5mg in healthy controls
  Arms: Normal
Drug: Dimebon — Dimebon 5mg in mild hepatic impairment patients
  Arms: Mild Hepatic Impairment
Drug: Dimebon — Dimebon 5mg in moderate hepatic impairment patients
  Arms: Moderate hepatic Impairment
Drug: Dimebon — Dimebon 5mg in Severe Hepatic Impairment
  Arms: Severe Hepatic Impairment

SUMMARY:
1. To compare the pharmacokinetics of Dimebon in subjects with mild and moderate hepatic impairment to subjects with normal hepatic function.
2. To assess the safety and tolerability of Dimebon in subjects with hepatic impairment and subjects with normal hepatic function.
3. To explore the pharmacokinetics of Dimebon in subjects with severely-impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (healthy is defined as the absence of clinically-relevant abnormalities identified by a detailed medical history, full physical examination, 12-lead ECG and clinical laboratory tests).
* Free of any medical or surgical conditions that might significantly interfere with gastrointestinal absorption, distribution, metabolism, or excretion of Dimebon.
* Demographically comparable to subjects with mild and moderate hepatic impairment.
* Subjects with hepatic impairment: Screening medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests performed within 28 days before the first dose of study medication, abnormal findings that are related to the subject's underlying condition are acceptable.
* Satisfy the criteria for Class A, B, or C of the modified Child-Pugh classification [Mild (Child-Pugh Scores 5-6 points), moderate (Child-Pugh Scores 7-9 points), and severe (Child-Pugh Scores >9 and <12 points)] within 14 days before the first dose of study medication.
* A diagnosis of hepatic impairment due to cirrhosis, not secondary to other diseases, which is confirmed and documented by medical history, physical examination, liver biopsy or hepatic ultrasound, CT scan or MRI.

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the trial:CYP2D6 PM genotype, as identified by screening genotyping.
* A known sensitivity to Dimebon.
* Exposure within the previous three months to a drug known to have a negative effect on skeletal muscle or reproductive organs.
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, active peptic ulcer within last 3 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax) | 1 day

SECONDARY OUTCOMES:
Safety (AEs, labs, ECG, vitals) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451018&StudyName=Study%20To%20Evaluate%20The%20Pharmacokinetics%2C%20Safety%2C%20And%20Tolerability%20Of%20Dimebon%20%5BPf-01913539%5D%20In%20Subjects%20With%20Hepatic%20Impairment%20And%20No